CLINICAL TRIAL: NCT02793843
Title: A Randomized Study Evaluating Preventive Role of Ondansetron Versus Ondansetron Plus Dexamethasone for Postoperative Side Effects of Intrathecal Morphine Injection in Patients Undergoing Elective C-section
Brief Title: Ondansetron vs Ondansetron Plus Dexamethasone for Relieving Intrathecal Morphine Side Effects After C-section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2432016
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Pruritus; Cesarean Section
MeSH Terms: conditions — Pruritus | interventions — Ondansetron; Dexamethasone; Calcium Dobesilate; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron (Active Comparator)
  Interventions: Drug: Ondansetron (Zofran); Other: Spinal anesthesia
- Ondansetron+ dexamethasone (Experimental)
  Interventions: Drug: Ondansetron (Zofran); Drug: Dexamethasone (Decadron); Other: Spinal anesthesia

INTERVENTIONS:
Drug: Ondansetron (Zofran) — Intravenous administration of 4 mg ondansetron 15 minutes before spinal anesthesia
Drug: Dexamethasone (Decadron) — Intravenous administration of 8 mg dexamethasone 15 minutes before spinal anesthesia
  Arms: Ondansetron+ dexamethasone
Other: Spinal anesthesia — Intrathecal anesthesia by 10 mg hyperbaric marcain, 5 mcg sufentanyl and 150 mcg morphine using 27 G spinal needle (27 G Quincke needle)

SUMMARY:
Background: Common adverse side effects related to the use of neuraxial opioids in the obstetric population include nausea, vomiting, and pruritus. Serotonin (5-HT3) receptor antagonists, in particular ondansetron, have been identified as possible antipruritic agents. It was reported that dexamethasone plus ondansetron is more effective than ondansetron for prevention of postoperative nausea and vomiting but no additional effect on treating pruritus.

Objectives: The purpose of this study is to compare the effect of prophylactic ondansetron versus ondansetron plus dexamethasone after cesarean section on pruritus and postoperative nausea and vomiting (PONV).

Methods: A prospective randomized double blind study that will be conducted between June 2016 and June 2017. Patients will be randomly allocated into two groups. The first group will receive 4 mg intravenous (IV) ondansetron while the other group will receive 4 mg IV ondansetron plus 8 mg dexamethasone.

DETAILED DESCRIPTION:
A prospective randomized double blind study will be conducted between June 2016 and June 2017. The sealed envelope technique will be used to randomly allocate females scheduled for elective cesarean section into two groups. After obtaining informed consent, all eligible patients will receive spinal anesthesia. The first group will receive 4 mg intravenous (IV) ondansetron with 2 ml saline while the other group will receive 4 mg IV ondansetron plus 8 mg (2 ml) dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status 1 and 2
* Scheduled for elective c-section surgery under spinal anesthesia

Exclusion Criteria:

* Patients with cardiac and psychological problems
* Patients who take sedatives or narcotics
* Patient who have allergy to study drugs

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06-15 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Pruritus assessed through questionnaire | 24 hours postoperatively

SECONDARY OUTCOMES:
Post operative nausea and vomiting assessed through questionnaire | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No